CLINICAL TRIAL: NCT06125145
Title: Tailored Geriatric Assessment and Promotores Pilot Feasibility Study
Brief Title: Geriatric Assessment and Promotores (GAP) Pilot Feasibility Study
Acronym: GAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1943526; 5K12CA138464 (NIH)
Record Dates: First submitted 2023-10-27; First posted 2023-11-09 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Colorectal Cancer; Prostate Cancer
Keywords: geriatrics; frailty; community health workers
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms; Frailty | interventions — Geriatric Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility Arm (Experimental): All enrolled participants will receive the pilot Geriatric Assessment and Promotora Coaching intervention.
  Interventions: Behavioral: Geriatric Assessment and Promotora Coaching

INTERVENTIONS:
Behavioral: Geriatric Assessment and Promotora Coaching — In Visit 1 the community health worker/promotora will assess frailty, cognition, polypharmacy, depression, symptom burden, and social support. In Visits 2 and 3 the community health worker will deliver interpersonal communication techniques to deliver the problem solving coaching format, leverage cultural congruence with clients, and provide social support to assist in adopting healthy behaviors.

SUMMARY:
The goal of this clinical trial is to test a new way to help older adults who have had cancer.

The researchers want to see if a program that assesses participants health and aging is achievable and makes a difference. A community health worker/promotora de salud will assess their health and provide coaching to help them feel better. This is important because older adults with cancer often have other health issues that are not addressed after completing treatment. The researchers want to make sure they get the care they need.

DETAILED DESCRIPTION:
The proposed study is a single arm feasibility study of a supportive care intervention. Phase is not applicable because this is not a drug trial. The study involves enrolling older adult non-metastatic cancer survivors between 1 month and 24 months after the completion of any definitive (e.g., curative intent) cancer treatment. The objective is to determine if a Community Health Worker (CHW)-led geriatric assessment and coaching intervention to assess geriatric syndromes is a feasible modality in community-dwelling older adult cancer survivors. The tailored assessment intervention (geriatric assessment and coaching) is hypothesized to potentially be a feasible process to monitor patients that would otherwise not access geriatric services after completing cancer treatment. Coping and social support are hypothesized mediators to the relationship between physical function and health outcomes (e.g., physical function, mental health), influenced by sociodemographic contextual factors. Implementation science concepts, such as acceptability and scalability will also be collected. The study CHW will perform the geriatric assessment and coaching components with each of the patients in the study. The assessment component of the bundle intervention involves screening for frailty and cognition, occurring prior to the coaching session. The CHW will conduct a more thorough geriatric assessment for polypharmacy, depression, symptom burden, and social support. In follow up visits after the geriatric assessment the CHW will deliver the coaching component (derived from the Problem Solving Coaching Model) to participants. Each of the intervention sessions will consist of 45-minute appointments with tailored feedback of the geriatric assessment domains, caregiver and family support, and navigation to additional palliative care resources at the study institution. The researchers developed the content in the tailored assessment intervention from preliminary work and thorough review of scientific literature.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65-90
2. Able to understand study procedures and to comply with them for the entire length of the study.
3. Diagnosis of Stage II-III breast, colorectal, or prostate cancer in within 1 to 24 months.
4. Completed course of definitive therapy within 12 months from enrollment into the study.
5. Proficient in English or Spanish
6. Reside within the UC Davis Health catchment area.
7. Has self-reported primary caregiver aged 21-90 years.

Exclusion Criteria:

1. Contraindication to any study-related procedure or assessment.
2. Patient is unable to independently deliver informed consent.
3. Patient screens positive for cognitive impairment (6CIT > 8)

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-19 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Describe the percentage of participants that complete 2 out of 3 study visits | 6 month
  Calculate percentage of participants that complete study compared to total enrolled (Goal: 65)

SECONDARY OUTCOMES:
Physical Function | Baseline to 6 month
  Patient-Reported Outcomes Measurement Information System [PROMIS] Physical Function
Depression, Anxiety, and Fatigue | Baseline to 6 month
  Patient-Reported Outcomes Measurement Information System [PROMIS] Depression, Anxiety, and Fatigue
Self-Efficacy | Baseline to 6 month
  Patient-Reported Outcomes Measurement Information System [PROMIS] Self-Efficacy
Emotional Support | Baseline to 6 month
  Patient-Reported Outcomes Measurement Information System [PROMIS] Emotional Support
Quality of Life in Elderly Cancer Patients | Baseline to 6 month
  European Organization for Research and Treatment of Cancer [EORTC] Quality of Life Questionnaire in the Elderly 14 item questionnaire [QLQ-ELD14]. Range 0 to 100, higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Fauer, PhD MS, Principal Investigator — UC Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No